CLINICAL TRIAL: NCT04065464
Title: TRACY - Track My Cycle
Acronym: TRACY
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Ava AG (Industry)
Responsible Party: Principal Investigator, Clare Barnett, MBBS (Hons) MPH, Director of Project Management, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2019_01
Record Dates: First submitted 2019-08-05; First posted 2019-08-22 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Fertility Monitor; Cycle Tracking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Ava Fertility Tracker — All women aged 18 to 40 years using Ava Fertility Tracker to track their cycles.

SUMMARY:
The primary aim of the pilot study is to collect data for the fine-tuning and evaluation of the Ava algorithm. Secondary outcomes are the estimation of the accuracy in detecting the fertility status of each cycle day.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 at the time of admission
* Not pregnant and no pregnancy wish during the pilot study period
* Have a regular sleep pattern (sleep at least four hours per night and not working nightshift)
* Have regular menstrual cycles

Exclusion Criteria:

* Pregnant at study admission
* Currently breastfeeding or have breastfed in the past 6 months before study admission
* Currently using hormonal contraception or hormonal medication
* Health-related conditions that may affect menstrual cycle length and variability (e.g. PCOS, menopause, thyroid dysfunction)
* Unable to understand study instructions and/or not able to understand English or German
* More than one international overseas travel per month
* Unwilling to sign the ICF.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: All women aged 18 to 40 years matching the eligibility criteria can be enrolled in the pilot study.
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Fine-tuning Ava algorithm | 5 months
  Number of days within a menstrual cycle that are correctly predicted as 'fertile' by the Ava algorithm.
  Number of study participants who have their 'fertile window' accurately predicted by the Ava AG app.

CONTACTS AND LOCATIONS:
Locations (1):
- ZEG Berlin, Mitte, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided